CLINICAL TRIAL: NCT04373434
Title: A Hybrid Effectiveness-Implementation Study on Weight Gain Prevention Among 2-1-1 Callers
Brief Title: Healthy Homes/Healthy Families (HH/HF) Intervention in 2-1-1 Callers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle C. Kegler, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00112359; CDC-IRB00112359 (Other: Centers for Disease Control and Prevention)
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Weight Change, Body
Keywords: Weight Gain Prevention; Cancer Prevention; Chronic Conditions; Obesity; Healthy Eating
MeSH Terms: conditions — Body Weight Changes; Chronic Disease; Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Homes/Healthy Families (HH/HF) Intervention (Experimental): Participants randomized to the HH/HF study intervention will work with a coach through phone calls and text messages for 12 weeks to set goals targeting home-based environmental determinants of dietary behaviors.
  Interventions: Behavioral: Health Homes/Healthy Families (HH/HF) Intervention
- Control (Active Comparator): Participants in the control condition will receive two mailings which focus on the same dietary outcomes as the HH/HF intervention but without the home environment emphasis.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Health Homes/Healthy Families (HH/HF) Intervention — The HH/HF Intervention involves coaching calls, text messages and intervention materials that are designed to increase behavioral capability, self-efficacy and behavioral intention to improve the home food environment for healthy eating and weight gain prevention. The intervention is delivered over a 12 week period.
  Arms: Healthy Homes/Healthy Families (HH/HF) Intervention
Behavioral: Control — Participants in the control condition will receive two mailings on healthy eating, the first from the "Dietary Guidelines For Americans 2015-2020, 8th Edition" and the second from "Choose MyPlate". Additionally, both mailings will include a food diary from the Centers for Disease Control and Prevention. Mailings will be sent to participants one and six-weeks post-baseline. These materials focus on the same dietary outcomes being targeted in the HH/HF intervention, but without the home environment emphasis. Control group participants will receive their home environment profile with a list of healthy actions upon completion of the study.
  Arms: Control

SUMMARY:
This trial will evaluate a healthy eating and weight gain prevention intervention for delivery through calls to the 2-1-1 number.

DETAILED DESCRIPTION:
It is now well-established that obesity and excess weight increase the risk of cancer (i.e., colorectal and post-menopausal breast cancer), as well as other chronic diseases including diabetes, stroke, coronary heart disease, and arthritis. The World Cancer Research Fund and the American Institute for Cancer Research state "maintenance of a healthy weight throughout life may be one of the most important ways to protect against cancer". Unfortunately, adults generally gain weight as they age.

Healthy Homes/Healthy Families (HH/HF) Intervention involves a tailored home environment profile and a health coach working with participants to select and implement a series of healthy actions to create a home environment more supportive of healthy eating and physical activity.

The Federal Communications Commission (FCC) designated 2-1-1 as the 3-digit number to call for information and referrals to social services and other assistance in the United States. This study will evaluate a healthy eating and weight gain prevention intervention for delivery through 2-1-1 calls.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* able to speak English
* self-report BMI of 20 and above

Exclusion Criteria:

* pregnant women
* only one member per household will be enrolled

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kegler, DrPH/MPH, Principal Investigator — Emory University
Locations (1):
- Emory University, Rollins School of Public Health, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results, after de-identification will be shared
Supporting Information: Study Protocol, SAP
Time Frame: Six months after publication of the primary results data will become available
Access Criteria: Researchers should send a methodologically sound proposal to mkegler@emory.edu. To gain access, requesters will need to sign a data access agreement. Upon approval, data will be shared via a secure website such as Box

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the United Way of Greater Atlanta 2-1-1, United Way of Central Georgia, United Way of the Chattahoochee Valley 2-1-1, and United Way of Southwest Georgia as part of a hybrid effectiveness implementation trial testing an adapted version of the Healthy Homes/Healthy Families healthy eating and weight gain prevention intervention. Participant enrollment began in September 2020, and final follow-up assessments were completed in December 2022.
Groups:
- Healthy Homes/Healthy Families (HH/HF) Intervention: Received a 12-week telephone-based healthy eating and weight gain prevention intervention, Healthy Homes/Healthy Families, that supports households in making changes in their home environment to promote healthy eating.
- Control: Received two mailings post baseline: first mailing included a food diary from the CDC, and healthy eating information from the Dietary Guidelines for Americans 2015-2020; Second mailing included the food diary and healthy eating information from Choose MyPlate
Period: Overall Study
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
Started | 255 | 257
Completed | 208 | 220
Not Completed | 47 | 37
Not completed — Lost to Follow-up | 37 | 32
Not completed — Refused at 9 months | 1 | 2
Not completed — Refused at 4 months | 7 | 3
Not completed — Excluded | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control | Total
Number analyzed (Participants) | 253 | 257 | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.2) | 43.0 (11.7) | 43.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 237 | 467
  Male | 23 | 20 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 250 | 250 | 500
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Some participants did not provide information for every baseline characteristic
  Participants
    Race: number analyzed (Participants) | 251 | 252 | 503
    Race: American Indian, Alaska Native Asian | 3 | 0 | 3
    Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0
    Race: Black or African American | 206 | 210 | 416
    Race: White | 31 | 21 | 52
    Race: More than one race | 8 | 14 | 22
    Race: Unknown or not reported | 3 | 7 | 10
Highest education [Count of Participants; unit: Participants]
  Less than high school | 20 | 24 | 44
  High school or GED | 66 | 86 | 152
  Some college/technical school | 103 | 91 | 194
  College graduate or higher | 64 | 56 | 120
Employment status [Count of Participants; unit: Participants]
  Employed | 143 | 138 | 281
  Not Employed | 110 | 119 | 229
Household income [Count of Participants; unit: Participants] — Population: Some participants did not provide information for every baseline characteristic.
  Participants
    number analyzed (Participants) | 241 | 246 | 487
    $10,000 and under | 66 | 70 | 136
    $10,001 - $20,000 | 57 | 67 | 124
    $20,001 - $35,000 | 55 | 67 | 122
    $35,001 - $50,000 | 35 | 27 | 62
    More than $50,000 | 28 | 15 | 43
Marital status [Count of Participants; unit: Participants]
  Married/living with partner | 63 | 49 | 112
  Widowed/separated/divorced | 62 | 56 | 118
  Not married | 128 | 152 | 280

OUTCOME MEASURES:

1. Primary Outcome: Change in United States Department of Agriculture (USDA) Healthy Eating Index (HEI)
Description: Description: The USDA HEI measures diet quality and is calculated from two telephone administered 24-hr dietary recalls (one weekday, one weekend day). The HEI evaluates foods with a scoring system using 13 components for different food groups and the key recommendations of the 2015-2020 "Dietary Guidelines for Americans." Scores range from 0 to 100 where a score of 100 is an ideal score indicating that a diet follows the key recommendations of the 2015-2020 "Dietary Guidelines for Americans" (higher scores indicate better diet quality).
Time Frame: Baseline, Month 4, Month 9
Population: Some participants were lost to follow-up. For the exact breakdown, kindly refer to the baseline characteristics above
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
Number analyzed (Participants) | 253 | 257
units on a scale
  Baseline | 51.0 (12.3) | 52.6 (12.9)
  Month 4 (Mean change from baseline ): number analyzed (Participants) | 219 | 211
  Month 4 (Mean change from baseline ) | 3.38 (14.45) | 0.92 (14.06)
  Month 9 (Mean change from baseline ): number analyzed (Participants) | 192 | 215
  Month 9 (Mean change from baseline ) | 2.74 (14.57) | -0.27 (14.10)

2. Secondary Outcome: Change in Kcal Per Day Intake
Description: Kcal per day will be calculated and recorded. The most recent version of the Automated Self-Administered 24-hour dietary recall (ASA24) program prompts for food description details and automatically codes and calculates nutrient intakes using the USDA Food and Nutrient Database for Dietary Studies. The average of one weekday and one weekend day will be used to estimate Kcal per day at each time point.
Time Frame: Baseline, Month 4, Month 9
Population: Some participants were lost to follow-up. For the exact breakdown, kindly refer to the baseline characteristics above.
Measure: Mean (Standard Deviation); unit: Kcal/day
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
Number analyzed (Participants) | 253 | 257
Kcal/day
  Baseline | 1736 (863.0) | 1718 (784.5)
  Month 4 (Mean change): number analyzed (Participants) | 219 | 211
  Month 4 (Mean change) | -206 (757) | -80 (743)
  Month 9 (Mean change): number analyzed (Participants) | 192 | 215
  Month 9 (Mean change) | -155 (908) | -93 (763)

3. Secondary Outcome: Change in Self-reported Weight
Description: Participants will self-report weight in pounds each time point
Time Frame: Baseline, Month 4, Month 9
Population: Some participants were lost to follow-up. For the exact breakdown, kindly refer to the baseline characteristics above
Measure: Mean (Standard Deviation); unit: weight in pounds (lbs)
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
Number analyzed (Participants) | 253 | 257
weight in pounds (lbs)
  Baseline | 202.3 (53.1) | 204.1 (51.9)
  Month 4 (Mean change from baseline ): number analyzed (Participants) | 220 | 213
  Month 4 (Mean change from baseline ) | -6.5 (21.74) | -2.9 (19.31)
  Month 9 (Mean change from baseline): number analyzed (Participants) | 203 | 220
  Month 9 (Mean change from baseline) | -4.5 (20.64) | -2.5 (21.17)

4. Secondary Outcome: Changes to Food Environment: UNHEALTHY SNACKS/FOODS INVENTORY, OF 8
Description: Participants were asked about unhealthy snacks and foods, ranging from 0 to 8, in each survey of the household food inventory. The higher the number the more unhealthy snacks/foods were reported
Time Frame: Baseline, Month 4, Month 9
Population: Some participants were lost to follow-up. For the exact breakdown, kindly refer to the baseline characteristics above
Measure: Mean (Standard Deviation); unit: number of unhealthy snacks in the home
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
Number analyzed (Participants) | 253 | 257
number of unhealthy snacks in the home
  Baseline | 4.29 (1.71) | 4.45 (1.72)
  Month 4: number analyzed (Participants) | 223 | 215
  Month 4 | -1.12 (2.05) | -0.18 (1.90)
  Month 9: number analyzed (Participants) | 207 | 221
  Month 9 | -0.75 (2.18) | -0.39 (2.10)

5. Secondary Outcome: Changes to Food Environment: PURCHASING FRUITS/VEGETABLES ≥1/WK
Description: A home environment survey assessed the frequency of shopping for or bringing home fruits and vegetables in the past month. Response options were 1=less than once per week, 2=once per week, or 3=more than once per week. Anyone who purchased fruits or vegetables at least once a week was scored as 1, while all others were scored as zero. Reporting includes the percentage of participants who scored 1, i.e., purchased fruits or vegetables at least once a week.
Time Frame: Baseline, Month 4, Month 9
Population: Some participants were lost to follow-up. For the exact breakdown, kindly refer to the baseline characteristics above
Measure: Number; unit: percentage of participants
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
Number analyzed (Participants) | 252 | 257
percentage of participants
  Baseline | 76.19 | 72.37
  Month 4: number analyzed (Participants) | 223 | 215
  Month 4 | 10.8 | 4.7
  Month 9: number analyzed (Participants) | 207 | 220
  Month 9 | 7.2 | 5.5

6. Secondary Outcome: Changes to Food Environment: HEALTHY FOOD PREPARATION
Description: Participants were asked about 16 food preparation methods and 3 food serving practices focused on portion control (e.g., use of smaller plates) in the past month. Response options were 1=never/rarely, 2=occasionally, 3=often, and 4=very often. Unhealthy food prep items were reverse-coded, and then all items were averaged. The higher the number, the more frequently healthy food preparation methods were used, and unhealthy food preparation methods were used less frequently
Time Frame: Baseline, Month 4, Month 9
Population: Some participants were lost to follow-up. For the exact breakdown, kindly refer to the baseline characteristics above
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
Number analyzed (Participants) | 253 | 257
units on a scale
  Baseline | 2.10 (0.44) | 2.12 (0.45)
  Month 4 (mean change from baseline): number analyzed (Participants) | 222 | 215
  Month 4 (mean change from baseline) | 0.21 (0.49) | -0.02 (0.40)
  Month 9 (mean change from baseline): number analyzed (Participants) | 207 | 221
  Month 9 (mean change from baseline) | 0.20 (0.48) | 0.05 (0.40)

7. Secondary Outcome: Changes to Food Environment: FAMILY MEALS FROM NONHOME SOURCES, DAYS IN PAST WEEK
Description: A home environment survey assessed non-home food sources. Participants were asked how many days in the last week (never, 1-7) they purchased a family meal from four non-home food sources (e.g. fast food, convenience store). The total score was calculated by adding the four types of meals with possible scores ranging from 0 to 28. A higher score indicated more family meals per week from non-home sources.
Time Frame: Baseline, Month 4, Month 9
Population: Some participants were lost to follow-up. For the exact breakdown, kindly refer to the baseline characteristics above
Measure: Mean (Standard Deviation); unit: meals per week
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
Number analyzed (Participants) | 253 | 257
meals per week
  Baseline | 3.27 (3.50) | 2.88 (2.94)
  Month 4 (mean change from baseline): number analyzed (Participants) | 223 | 214
  Month 4 (mean change from baseline) | -0.59 (3.59) | -0.12 (3.02)
  Month 9 (mean change from baseline): number analyzed (Participants) | 207 | 221
  Month 9 (mean change from baseline) | -0.67 (4.30) | -0.01 (3.44)

8. Secondary Outcome: Changes to Food Environment: Family Eating and TV
Description: A home environment survey included two items on meals/snacks eaten with the television on. Response options ranged: 1=never/rarely, 2=occasionally, 3=often, 4=very often. The score was calculated as the mean of both items. A higher score indicates more frequently eaten meals and snacks with the television on.
Time Frame: Baseline, Month 4, Month 9
Population: Some participants were lost to follow-up. For the exact breakdown, kindly refer to the baseline characteristics above
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
Number analyzed (Participants) | 253 | 257
units on a scale
  Baseline | 2.65 (1.02) | 2.58 (1.09)
  Month 4 (mean change from baseline): number analyzed (Participants) | 223 | 215
  Month 4 (mean change from baseline) | -0.55 (1.08) | -0.16 (1.03)
  Month 9 (mean change from baseline): number analyzed (Participants) | 207 | 221
  Month 9 (mean change from baseline) | -0.45 (1.10) | -0.17 (1.04)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Month 12
Arm/Group | Healthy Homes/Healthy Families (HH/HF) Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/257
Serious Adverse Events (participants affected / at risk) | 0/253 | 0/257
Other Adverse Events (participants affected / at risk) | 0/253 | 0/257

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT04373434/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT04373434/ICF_000.pdf